CLINICAL TRIAL: NCT01355471
Title: A Multicenter, Randomized Double-Blind, Vehicle-Controlled, Parallel Group Study to Demonstrate the Efficacy and Safety of CD07805/47 Gel Applied Topically Once Daily in Subjects With Moderate to Severe Facial Erythema Associated With Rosacea
Brief Title: Phase 3 Efficacy and Safety Study of CD07805/47 Topical Gel in Subjects With Facial Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.18141
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2013-09

CONDITIONS: Rosacea
Keywords: rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD07805/47 gel (Experimental)
  Interventions: Drug: CD07805/47 Gel
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CD07805/47 Gel — applied topically once daily
  Arms: CD07805/47 gel
Drug: Placebo — applied topically once daily
  Arms: Placebo

SUMMARY:
This is a Phase 3 efficacy and safety study of CD07805/47 topical gel in subjects with facial erythema associated with rosacea. The study hypothesis is that CD07805/47 gel, applied topically once daily is more efficacious than vehicle and provides an acceptable safety profile in the treatment of facial erythema associated with rosacea.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female who is at least 18 years of age or older.
2. A clinical diagnosis of facial rosacea.
3. A Clinician Erythema Assessment (CEA) score of greater than or equal to 3 at Screening and at Baseline/Day 1 (prior to the study drug application).
4. A Patient Self Assessment (PSA) score of greater than or equal to 3 at Screening and at Baseline/Day 1 (prior to the study drug application).

Key Exclusion Criteria:

1. Particular forms of rosacea (rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, acute lupus erythematosus, or actinic telangiectasia.
2. Presence of three (3) or more facial inflammatory lesions of rosacea.
3. Current treatment with monoamine oxidase (MAO) inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, or alpha agonists.
4. Less than 3 months stable dose treatment with tricyclic antidepressants, cardiac glycosides, beta blockers or other antihypertensive agents.
5. Current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 293 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Chair — Galderma R&D; Kirk Barber, MD, Principal Investigator — Kirk Barber Research Inc.; Leslie Baumann, MD, Principal Investigator — Baumann Cosmetic and Research Institute; Fran Cook-Bolden, MD, Principal Investigator — Skin Specialty Dermatology; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists PSC; Steven Grekin, DO, Principal Investigator — Grekin Skin Institute; Wayne Gulliver, MD, Principal Investigator — Newlab Clinical Research Inc.; Robert Haber, MD, Principal Investigator — Haber Dermatology & Cosmetic Surgery; Michael Heffernan, MD, Principal Investigator — Central Dermatology; Terry Jones, MD, Principal Investigator — J&S Studies Inc.; Ian Landells, MD, Principal Investigator — Nexus Clinical Research; Mark Ling, MD, Principal Investigator — MedaPhase, Inc.; Phoebe Rich, MD, Principal Investigator — Oregon Dermatology and Research Center; Dow Stough, MD, Principal Investigator — Burke Pharmaceutical Research; William Werschler, MD, Principal Investigator — Premier Clinical Research; Patricia Westmoreland, MD, Principal Investigator — Palmetto Clinical Trials Services, LLC
Locations (15):
- United States (12):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Baumann Cosmetic and Research Institute, Miami Beach, Florida
  - MedaPhase, Inc., Newnan, Georgia
  - Dermatology Specialists Research, Louisville, Kentucky
  - Grekin Skin Institute, Warren, Michigan
  - Central Dermatology PC, St Louis, Missouri
  - Skin Specialty Dermatology, New York, New York
  - Haber Dermatology & Cosmetic Surgery, South Euclid, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - J&S Studies Inc., College Station, Texas
  - Premier Clinical Research, Spokane, Washington
- Canada (3):
  - Kirk Barber Research Inc., Calgary, Alberta
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Newlab Clinical Research Inc., St. John's, Newfoundland and Labrador

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CD07805/47 Gel | Placebo
Started | 148 | 145
Completed | 141 | 142
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD07805/47 Gel | Placebo | Total
Number analyzed (Participants) | 148 | 145 | 293
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 136 | 134 | 270
  >=65 years | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11.94) | 46.5 (12.10) | 47.5 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 108 | 213
  Male | 43 | 37 | 80
Region of Enrollment [Number; unit: participants]
  United States | 140 | 138 | 278
  Canada | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Composite Success
Description: Composite Success is defined as 2-grade improvement on both Clinician Erythema Assessment (CEA) and Patient Self Assessment(PSA).
Time Frame: Day 29
Population: Intent-to-Treat (ITT) population(i.e. Hours 3,6,9,12)
Measure: Number; unit: participants
Arm/Group | CD07805/47 Gel | Placebo
Number analyzed (Participants) | 142 | 142
participants
  Day 29/ Hour 3 | 36 | 13
  Day 29 / Hour 6 | 36 | 13
  Day 29 / Hour 9 | 25 | 15
  Day 29 / Hour 12 | 30 | 14
Statistical Analysis 1: Comparison: CD07805/47 Gel vs Placebo; Test type: Superiority or Other; p < 0.001, GEE: Logit link function; Generalized Estimation Equation (GEE) methods with Logit link function and marginal expectation model

ADVERSE EVENTS:
Arm/Group | CD07805/47 Gel | Placebo
Serious Adverse Events (participants affected / at risk) | 1/148 | 0/145
Other Adverse Events (participants affected / at risk) | 0/148 | 0/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CD07805/47 Gel (N=148) | Placebo (N=145)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days